CLINICAL TRIAL: NCT05569018
Title: Efficacy of a Group Treatment Based on Transdiagnostic Perspective for Emotional Disorders and Applied in Blended Format: a Randomized Controlled Trial.
Brief Title: Efficacy of a Transdiagnostic Group Treatment for Emotional Disorders Applied in Blended Format: a Controlled Study.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UJaumeI_Transd_Group_Blended_2
Record Dates: First submitted 2022-07-14; First posted 2022-10-06 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Anxiety Disorders; Depressive Disorders
Keywords: Cognitive-Behavioral Therapy; Transdiagnostic CBT; Blended CBT; Group CBT; Emotional disorders
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blended group transversal protocol (BLGr-TP) (Experimental): Treatment protocol based on the transdiagnostic perspective administered in blended (face-to-face + online) and group format. It consists of the following components: Psychoeducation about emotional disorders and emotion regulation; Motivation for change; Psychoeducation about emotions; Awareness of emotional experiences; Promotion of cognitive flexibility; Psychoeducation and awareness of avoidance strategies that maintain emotional problems; Interoceptive exposure: exposure to physical sensations; Situational and emotional exposure; Learning to move on; Learning to enjoy; Learning to live; Living and learning; Relapse prevention.
  Interventions: Behavioral: Blended group transversal protocol (BLGr-TP)
- Face-to-face group transversal protocol (FFGr-TP) (Active Comparator): Treatment protocol based on the transdiagnostic perspective administered in traditional (face-to-face) group format. It consists of the following components: Psychoeducation about emotional disorders and emotion regulation; Motivation for change; Psychoeducation about emotions; Awareness of emotional experiences; Promotion of cognitive flexibility; Psychoeducation and awareness of avoidance strategies that maintain emotional problems; Interoceptive exposure: exposure to physical sensations; Situational and emotional exposure; Learning to move on; Learning to enjoy; Learning to live; Living and learning; Relapse prevention.
  Interventions: Behavioral: Face-to-face group transversal protocol (FFGr-TP)

INTERVENTIONS:
Behavioral: Blended group transversal protocol (BLGr-TP) — It will consist in the administration of a transdiagnostic treatment protocol composed by 16 modules focused on regulating both negative and positive affect. The intervention will be administered over a 16-week period. Face-to-face group sessions will be combined with autonomous work of patients through a web platform where they will find the contents of the program. The groups will have 6-10 patients, who will attend a total of 8 face-to-face sessions of 2 hours long each one. The online part of the treatment (self-applied Online Transversal Protocol) will consist in working the contents exposed in the face-to-face sessions during between-sessions period (2 weeks). It is an interactive program with multimedia elements (videos, images,…) that allows people to perform the modules from home and at their own pace. In addition, the program is characterized by its ease of use, presenting an agile navigation.
  Other Names: BLGr-TP
  Arms: Blended group transversal protocol (BLGr-TP)
Behavioral: Face-to-face group transversal protocol (FFGr-TP) — It will consist in the administration of the transdiagnostic treatment protocol through the 16 modules focused on regulating both negative and positive affect. The intervention will be carried out in face-to-face group format and it will be administered during a 16-week period. The groups will have between 6 to 10 patients, who will attend a total of 16 face-to-face sessions of 2 hours long each one. During between-sessions period (1 week), patients will work the content of the modules exposed in the face-to-face sessions through tasks for home (traditional paper format).
  Other Names: FFGr-TP
  Arms: Face-to-face group transversal protocol (FFGr-TP)

SUMMARY:
This study will consist in a randomized controlled clinical trial (RCT) to test the efficacy of a blended group transversal protocol (BLGr-TP) compared to a face-to-face group transversal protocol (FFGr-TP).

The main aims of the study are the following:

* To analyze the differential efficacy of the BLGr-TP versus the FFGr-TP for the treatment of emotional disorders in aspects of clinical measures, as well as in terms of retention and dropout rate and adherence.
* To analyze the differential acceptability of the BLGr-TP versus the FFGr-TP for the treatment of emotional disorders.

In addition, it is intended to carry out a study of mediators and moderators of the efficacy of both interventions.

The established hypotheses in relation to the main goals are:

* Both treatment modalities (FFGr-TP and BLGr-TP) will achieve improvements in the symptoms of emotional disorders, reflected in the scores of the clinical measures.
* The BLGr-TP will show equivalent efficacy to the FFGr-TP.
* The BLGr-TP will show an acceptability comparable to the face-to-face protocol. Both modalities will be well valued by the participants.
* In both treatment modalities, the changes achieved are expected to be maintained over time (3, 6 and 12 months).

DETAILED DESCRIPTION:
Emotional disorders (ED) are among the most common and most disabling psychological disorders. They involve important costs and a high comorbidity between them. A large number of evidence-based treatment programs (EBT) has shown to be effective; however, there is a difficulty regarding their dissemination, being that it is difficult to train clinicians in the different protocols for different disorders, and a difficulty in the management of patients with comorbidity. The transdiagnostic approach and the incorporation of technologies for the administration of the based-Internet treatments can help to overcome these barriers. In this context, blended treatments, that combine face-to-face therapy with online therapy, are gaining prominence, because they exhibit advantages over traditional intervention and over treatments totally self-administered throughout Internet. Otherwise, the application of treatments in group format also allows to provide EBTs at a lower cost, so that both blended format and group format constitute strategies that allow improve the cost-effectiveness binomial. To our knowledge, no studies that integrate blended with group format for apply a transdiagnostic protocol for ED have been published.

This study will be a two-arm, parallel-group, randomized controlled clinical trial (RCT) in which participants will be randomly assigned to one of two conditions: 1) Face-to-face group transversal protocol (FFGr-TP) and 2) Blended group transversal protocol (BLGr-TP). To carry it out, a total of 144 patients will be needed. Randomization will be stratified by primary diagnosis. Block randomization will be performed within each stratum to ensure that all major diagnoses are equally represented under all conditions. In this trial there will be five evaluation moments: pre-treatment, post-treatment and follow-up at 3, at 6 and at 12 months. During the treatment administration, two messages of support (an email and a SMS) per week will be sent to participants.

The study will be carried out following national and international standards (Declaration of Helsinki and Tokyo, and Declaration of Madrid of the World Psychiatric Association) and has been submitted to the approval of the Research Ethics Committee of the Universitat Jaume I. Participants will be adult people who contact with the Psychological Assistance Service (PAS) of the Universitat Jaume I or who write at email enabled for the study. All participants will be volunteers and they will give their informed consent to participate in the study. The confidentiality and rights of the subjects included in the study will be guaranteed in accordance with the provisions of Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of the digital rights (LOPDgdd), which adapts Spanish legislation to the General Data Protection Regulation of the European Union (RGPD).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or more.
* DSM-5 (APA, 1013) diagnostic criteria for emotional disorder (panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder, major depressive disorder, dysthymia, obsessive-compulsive disorder, non-specified anxiety disorder, non-specified depressive disorder).
* Good understanding of Spanish.
* Access to the Internet and email address.
* Informed consent to participate.

Exclusion Criteria:

* Diagnosis of a severe mental disorder (psychotic disorder, bipolar disorder, substance and/or alcohol dependence).
* High risk of suicide.
* Having a serious medical illness or other condition that prevents treatment from being carried out.
* Receiving another psychological treatment during the study period.
* Changes and/or increases in pharmacological treatment during the study period (a decrease is accepted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in the Overall Anxiety Severity and Impairment Scale (OASIS) (Campbell-Sills et al., 2009; González-Robles et al., 2018) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-modules (throughout the treatment), post-treatment (4 months), follow-up (7, 10 and 16 months)
  The OASIS is a 5-item self-report scale that evaluates the frequency and severity of anxiety symptoms, the functional impairment related to these symptoms (i.e. school, work, home, or social impairment), and behavioral avoidance. Each item instructs respondents to endorse one of five responses that best describes their experiences over the past week. Response items are coded from 0 to 4, added together to obtain a total score ranging from 0 to 20. Previous studies have shown good internal consistency (α = 0.80), test-retest reliability, and convergent and discriminant validity. The Spanish version has shown good internal consistency (α = 0.86), and convergent and discriminant validity.
Change in the Overall Depression Severity and Impairment Scale (ODSIS) (Bentley et al., 2014; Mira et al., 2019) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-modules (throughout the treatment), post-treatment (4 months), follow-up (7, 10 and 16 months)
  The ODSIS is a brief self-reported scale with 5 items that assess the severity and functional impairment associated with depressive symptoms. Items are coded on a 5-point scale (0-4). The sum of the scores is used to obtain the total score, which can be a maximum of 20. The measure has shown excellent internal consistency (α = 0.94 in an outpatient sample, 0.92 in a community sample, and 0.91 in a student sample) and good convergent/discriminant validity. The Spanish validation has excellent internal consistency (α = 0.93), as well as convergent and discriminant validity.

SECONDARY OUTCOMES:
Change in the Positive and Negative Affect Schedule (PANAS) (Watson, Clark & Tellegen, 1988; Sandín et al., 1999; Díaz-García et al., 2020) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-modules (throughout the treatment), post-treatment (4 months), follow-up (7, 10 and 16 months)
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). It contains 10 descriptors evaluating PA (e.g., "enthusiastic", "inspired", "proud") and 10 others assessing NA (e.g., "scared", "irritable", "guilty"). The range for each scale (10 items on each) is from 10 to 50, and the patient has to answer how he or she usually feels regarding each of these emotions. The scale showed excellent internal consistency (α between .84 and .90) and convergent and discriminant validity. The Spanish version has demonstrated good to excellent internal consistency (α = .89 and .91 for PA and NA in women, respectively, and α = .87 and .89 for PA and NA in men, respectively) in college students.
Change in the Difficulties in Emotion Regulation Scale (DERS) (Gratz & Roemer, 2004; Hervás & Jódar, 2008) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-treatment (4 months), follow-up (7, 10 and 16 months)
  The DERS is a self-report scale that assesses different clinically relevant aspects of maladaptive emotional regulation and the main difficulties that may arise in the processing of emotions. In the Spanish adaptation of the scale, the factorial analysis showed five interpretable factors, one less than the original scale: Emotional lack of control (Impulsivity and No strategies of the original scale), Emotional rejection (No acceptance), Everyday interference (No goals), Emotional inattention (No awareness) and Emotional confusion (No clarity). The Spanish validation consists of 28 items with a 5-point Likert scale, being 1 = Almost never (0-10% of the time) and 5 = Almost always (90-100% of the time). The adapted scale has good psychometric properties: internal consistency of 0.93, test-retest reliability of 0.74 and good convergent and incremental validity.
Change in the NEO-Five Factor Inventory (NEO-FFI) (Costa & McCrae, 1992; Robins, Fraley, Roberts & Trzesniewski, 2001; Aluja, García, Rossier & García, 2005) at pre-treatment, post-treatmen,t and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-treatment (4 months), follow-up (7, 10 and 16 months)
  The NEO-FFI is the short version of the NEO-PI-R, designed to assess the five personality dimensions through 60 items. In this study, only the subscales of neuroticism and extraversion are used. Each scale contained 12 items with a five-point Likert response format. Two-week retest reliability is uniformly high, ranging from 0.86 to 0.90 for the five scales, and internal consistency ranges from 0.68 to 0.86. The Spanish version of the NEO-FFI has been found to be appropriate.
Change in the Quality of Life Index (QLI) (Mezzich, Cohen, Ruiperez, Benzato & Zapata-Vega, 2011; Mezzich et al., 2000) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-treatment (4 months), follow-up (7, 10 and 16 months)
  The QLI is a self-report questionnaire that consists of 10 items aimed at assessing quality of life in ten areas: psychological well-being, physical well-being, emotional and social support, interpersonal functioning, selfcare and independent functioning, community and service support, occupational functioning, self-realization, spiritual satisfaction, and an overall assessment of quality of life. The Spanish version of the QLI has shown good internal consistency and test-retest reliability in previous studies.
Change in the Work and Social Adjustment Scale (WSAS) (Echezarraga et al., 2018; Mundt et al., 2002) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-treatment (4 months), follow-up (7, 10 and 16 months)
  The WSAS is a 5-item scale that evaluates the degree of interference associated with the patients' symptoms in the following five domains: work, home management, private leisure, social leisure, and family relationships. Items are coded on a scale from 0 (not at all) to 8 (very severely), and higher scores are indicative of greater interference in the different areas. The scale has shown good to excellent internal consistency (α = 0.70 to 0.94), test-retest reliability, and sensitivity to change. The Spanish version has demonstrated excellent internal consistency and good concurrent validity.
Change on the Multidimensional Emotional Disorders Inventory (MEDI) (Rosellini & Brown, 2019; Osma et al., 2023) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-treatment (4 months), follow-up (7, 10 and 16 months)
  It is a self-report questionnaire that assesses nine transdiagnostic dimensions (Neurotic Temperament, Positive Temperament, Depressive Mood, Autonomic Arousal, Somatic Anxiety, Social Anxiety, Intrusive Thoughts, Traumatic Re-experiencing and Avoidance). It consists of a 49-item scale with a 9-point Likert-type response (from 0 = "It is not characteristic of me" to 8 = "Totally characteristic of me"). The Spanish validation shows good psychometric properties and strong internal consistency indices (α = 0.66 to 0.91).
Change on the General Self-Efficacy Scale (GSES) (Baessler y Schwarzer, 1996; Sanjuán et al., 2000) at pre-treatment, post-treatment, and at 3-, 6- and 12-month follow-up. | Pre-treatment, post-modules (throughout the treatment), post-treatment (4 months), follow-up (7, 10 and 16 months)
  It assesses the stable feeling of personal competence to effectively handle a wide variety of stressful situations. It consists of 10 items with 10-point Likert-type scales, so that subjects' scores can range from 10 to 100.
Change on the Modulate Subscale of the S-DERS (Lavender et al., 2017). | Throughout the treatment (post-modules measure)
  The S-DERS is a measure of difficulties in state emotional regulation, to assess momentary emotional regulation. Factor 2 (Modulate) includes items that reflect difficulties in responding emotionally and behaviorally in the moment, and was labeled as Limited Ability to Modulate Current Emotional and Behavioral Responses. This factor conceptually overlaps with the Strategies, Impulse, and Goals subscales of the original trait DERS, combining difficulties in modulating both emotions and behavioral responses to emotions into a single state scale. The Modulate subscale demonstrated adequate to excellent internal consistency (α=0.85). Regarding validity, the Modulate subscale was positively associated with measures of experiential avoidance, with measures of substance use problems, and with emotional reactivity.

OTHER OUTCOMES:
Score on the Expectations scale (adapted from Borkovec & Nau, 1972). | Pre-treatment
  This scale is made up of five items, rated on a scale from 0 (nothing at all) to 10 (completely), that cover how logical the treatment seems to be, to what extent it could satisfy the patient, whether it could be recommended to a person with the same problem, whether it could be used to treat other psychological problems, and its usefulness for the patient's problem. The Expectation Scale is applied once the treatment rationale has been explained. Its aim is to measure subjective patient expectations about this treatment.
Score on the Opinion scale (adapted from Borkovec & Nau, 1972). | Post-treatment (4 months)
  This scale is made up of five items, rated on a scale from 0 (nothing at all) to 10 (completely), that cover how logical the treatment seems to be, to what extent it could satisfy the patient, whether it could be recommended to a person with the same problem, whether it could be used to treat other psychological problems, and its usefulness for the patient's problem. The Opinion Scale is administered when the patient has completed the treatment, and its aim is to assess satisfaction with this treatment.
Score on the System Usability Scale (SUS) (Bangor, Kortum & Miller, 2008; Brooke, 1996). | Post-module 1 (1 week), Post-treatment (4 months)
  The SUS is applied in order to assess the usability of a service or product and the acceptance of technology by the people who use it. The SUS is a simple, ten-item scale that indicates the degree of agreement or disagreement with the statements on a 5-point scale (1 = strongly disagree, 5 = strongly agree). The final score is obtained by adding the scores on each item and multiplying the result by 2.5. Scores range from 0 to 100, where higher scores indicate better usability.
Score on the Working Alliance Inventory short format (WAI-S) (Corbella et al., 2011). | Post-module 3 (3 weeks)
  The WAI-S maintains the three subscales of the WAI and consists of 12 items to be answered on a 7-point Likert scale where the lower polarity is "never" and the upper polarity is "always". Each subscale (Goals, Tasks and Bond) is evaluated by 4 items. Thus, the total score of the WAI-S can range from 12 to 84 points.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Díaz-García, Dr., Principal Investigator — University of Zaragoza, Teruel Campus; Noelia Jiménez-Orenga, PhD student, Principal Investigator — Jaume I University, Castellón, Spain; Juana María Bretón-López, Dr., Principal Investigator — Jaume I University, Castellón, Spain; Azucena García-Palacios, Dr., Study Director — Jaume I University, Castellón, Spain

REFERENCES:
- [Background] Aluja, A., García, O., Rossier, J., et al. (2005). Comparison of the NEO-FFI, the NEOFFI-R and an alternative short version of the NEO-PI-R (NEO-60) in Swiss and Spanish samples. Pers Individ Dif, 38(3), 591-604.
- [Background] Andrews G, Basu A, Cuijpers P, Craske MG, McEvoy P, English CL, Newby JM. Computer therapy for the anxiety and depression disorders is effective, acceptable and practical health care: An updated meta-analysis. J Anxiety Disord. 2018 Apr;55:70-78. doi: 10.1016/j.janxdis.2018.01.001. Epub 2018 Feb 1. PMID 29422409
- [Background] Bangor, A., Kortum, P.T y Miller, J.T. (2008). An empirical evaluation of the System Usability Scale. International Journal of Human-Computer Interaction, 24(6), 574-594. https://doi.org/10.1080/10447310802205776
- [Background] Bentley KH, Gallagher MW, Carl JR, Barlow DH. Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess. 2014 Sep;26(3):815-830. doi: 10.1037/a0036216. Epub 2014 Apr 7. PMID 24708078
- [Background] Borkovec, T. D., & Nau, S. D. (1972). Credibility of analogue therapy rationales. Journal of behavior therapy and experimental psychiatry, 3(4), 257-260.
- [Background] Brooke, J. (1996). SUS: A 'Quick and Dirty' Usability Scale. In P. W. Jordan, B. Thomas, I. L. McClelland & B. Weerdmeester (Eds.), Usability Evaluation in Industry. London, England: CRC Press.
- [Background] Brown TA, Barlow DH. A proposal for a dimensional classification system based on the shared features of the DSM-IV anxiety and mood disorders: implications for assessment and treatment. Psychol Assess. 2009 Sep;21(3):256-71. doi: 10.1037/a0016608. PMID 19719339
- [Background] Campbell-Sills L, Norman SB, Craske MG, Sullivan G, Lang AJ, Chavira DA, Bystritsky A, Sherbourne C, Roy-Byrne P, Stein MB. Validation of a brief measure of anxiety-related severity and impairment: the Overall Anxiety Severity and Impairment Scale (OASIS). J Affect Disord. 2009 Jan;112(1-3):92-101. doi: 10.1016/j.jad.2008.03.014. Epub 2008 May 16. PMID 18486238
- [Background] Carlbring P, Andersson G, Cuijpers P, Riper H, Hedman-Lagerlof E. Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: an updated systematic review and meta-analysis. Cogn Behav Ther. 2018 Jan;47(1):1-18. doi: 10.1080/16506073.2017.1401115. Epub 2017 Dec 7. PMID 29215315
- [Background] Costa, P. T. & McCrae, R. R. (1992). Normal personality assessment in clinical practice: the NEO personality inventory. Psychol. Assess., 4(1), 5-13.
- [Background] Diaz-Garcia A, Gonzalez-Robles A, Mor S, Mira A, Quero S, Garcia-Palacios A, Banos RM, Botella C. Positive and Negative Affect Schedule (PANAS): psychometric properties of the online Spanish version in a clinical sample with emotional disorders. BMC Psychiatry. 2020 Feb 10;20(1):56. doi: 10.1186/s12888-020-2472-1. PMID 32039720
- [Background] Diaz-Garcia A, Gonzalez-Robles A, Garcia-Palacios A, Fernandez-Felipe I, Tur C, Castilla D, Botella C. Blended transdiagnostic group CBT for emotional disorders: A feasibility trial protocol. Internet Interv. 2021 Jan 7;23:100363. doi: 10.1016/j.invent.2021.100363. eCollection 2021 Mar. PMID 33520670
- [Background] Echezarraga A, Calvete E, Las Hayas C. Validation of the Spanish Version of the Work and Social Adjustment Scale in a Sample of Individuals With Bipolar Disorder. J Psychosoc Nurs Ment Health Serv. 2019 May 1;57(5):44-51. doi: 10.3928/02793695-20181128-02. Epub 2018 Dec 4. PMID 30508459
- [Background] Gonzalez-Robles A, Mira A, Miguel C, Molinari G, Diaz-Garcia A, Garcia-Palacios A, Breton-Lopez JM, Quero S, Banos RM, Botella C. A brief online transdiagnostic measure: Psychometric properties of the Overall Anxiety Severity and Impairment Scale (OASIS) among Spanish patients with emotional disorders. PLoS One. 2018 Nov 1;13(11):e0206516. doi: 10.1371/journal.pone.0206516. eCollection 2018. PMID 30383797
- [Background] Gratz, K. L., & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54.
- [Background] Hervás, G. & Jódar, R. Adaptación al castellano de la Escala de Dificultades en la Regulación Emocional. Clínica y Salud, 19(2), 139-156.
- [Background] Kobak KA, Mundt JC, Kennard B. Integrating technology into cognitive behavior therapy for adolescent depression: a pilot study. Ann Gen Psychiatry. 2015 Nov 3;14:37. doi: 10.1186/s12991-015-0077-8. eCollection 2015. PMID 26535048
- [Background] Kooistra LC, Wiersma JE, Ruwaard J, van Oppen P, Smit F, Lokkerbol J, Cuijpers P, Riper H. Blended vs. face-to-face cognitive behavioural treatment for major depression in specialized mental health care: study protocol of a randomized controlled cost-effectiveness trial. BMC Psychiatry. 2014 Oct 18;14:290. doi: 10.1186/s12888-014-0290-z. PMID 25326035
- [Background] Mezzich JE, Cohen NL, Ruiperez MA, Banzato CE, Zapata-Vega MI. The Multicultural Quality of Life Index: presentation and validation. J Eval Clin Pract. 2011 Apr;17(2):357-64. doi: 10.1111/j.1365-2753.2010.01609.x. Epub 2011 Jan 5. PMID 21208350
- [Background] Mezzich JE, Ruiperez MA, Perez C, Yoon G, Liu J, Mahmud S. The Spanish version of the quality of life index: presentation and validation. J Nerv Ment Dis. 2000 May;188(5):301-5. doi: 10.1097/00005053-200005000-00008. PMID 10830568
- [Background] Mira A, Gonzalez-Robles A, Molinari G, Miguel C, Diaz-Garcia A, Breton-Lopez J, Garcia-Palacios A, Quero S, Banos R, Botella C. Capturing the Severity and Impairment Associated With Depression: The Overall Depression Severity and Impairment Scale (ODSIS) Validation in a Spanish Clinical Sample. Front Psychiatry. 2019 Apr 9;10:180. doi: 10.3389/fpsyt.2019.00180. eCollection 2019. PMID 31024352
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Robins RW, Fraley RC, Roberts BW, Trzesniewski KH. A longitudinal study of personality change in young adulthood. J Pers. 2001 Aug;69(4):617-40. doi: 10.1111/1467-6494.694157. PMID 11497032
- [Background] Sandín, B., Chorot, P., Lostao, L., et al. (1999). Escalas PANAS de afecto positivo y negativo: validacion factorial y convergencia transcultural. Psicothema, 11(1), 37-51.
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Rosellini AJ, Brown TA. The Multidimensional Emotional Disorder Inventory (MEDI): Assessing transdiagnostic dimensions to validate a profile approach to emotional disorder classification. Psychol Assess. 2019 Jan;31(1):59-72. doi: 10.1037/pas0000649. Epub 2018 Aug 30. PMID 30160498
- [Background] Osma J, Martinez-Loredo V, Quilez-Orden A, Peris-Baquero O, Ferreres-Galan V, Prado-Abril J, Torres-Alfosea MA, Rosellini AJ. Multidimensional emotional disorders inventory: Reliability and validity in a Spanish clinical sample. J Affect Disord. 2023 Jan 1;320:65-73. doi: 10.1016/j.jad.2022.09.140. Epub 2022 Sep 29. PMID 36183816
- [Background] Baessler, J. & Schwarcer, R. (1996). Evaluación de la autoeficacia: Adaptación española de la escala de Autoeficacia General. Ansiedad y Estrés, 2, 1-8.
- [Background] Sanjuán, P., Pérez, A., Bermúdez, J., 2000. Escala de autoeficacia general: Datos psicométricos de la adaptación para población española. Psicothema 12.
- [Background] Corbella, S., Botella, L., Gómez, A.M., Herrero, O., Pacheco, M., 2011. Características psicométricas de la versión española del Working Alliance Inventory-Short (WAI-S). Anales de psicología, 27(2), 298-301.
- [Background] Lavender JM, Tull MT, DiLillo D, Messman-Moore T, Gratz KL. Development and Validation of a State-Based Measure of Emotion Dysregulation. Assessment. 2017 Mar;24(2):197-209. doi: 10.1177/1073191115601218. Epub 2016 Jul 27. PMID 26297011
- [Derived] Jimenez-Orenga N, Diaz-Garcia A, Garcia-Palacios A, Breton-Lopez J. Effectiveness of a blended group transdiagnostic treatment for emotional disorders: Study protocol for a randomized controlled trial. Internet Interv. 2024 Jul 30;37:100761. doi: 10.1016/j.invent.2024.100761. eCollection 2024 Sep. PMID 39188940
- See also: Web platform of self-applied treatment — http://psicologiaytecnologia.labpsitec.es/